CLINICAL TRIAL: NCT01828840
Title: A Prospective Double Blind Randomized Comparison of Methadone, Fentanyl, and Morphine for Post-laparotomy Epidural Analgesia.
Brief Title: A Prospective Comparison of Methadone, Fentanyl, and Morphine for Post-laparotomy Epidural Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0080-10-HMO
Record Dates: First submitted 2013-01-13; First posted 2013-04-11 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2016-03

CONDITIONS: Post Laparotomy Pain Treatment
Keywords: morphine; fentanyl; methadone; epidural; intravenous; pain; analgesia
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- morphine, epidural (Active Comparator): Epidurally administrated morphine
  Interventions: Drug: epidural morphine via PCEA
- fentanyl, epidural (Active Comparator): epidurally administrated fentanyl
  Interventions: Drug: epidural fentanyl via PCEA
- methadone, epidural (Active Comparator): epidurally administrated methadone
  Interventions: Drug: epidural methadone via PCEA
- morphine, intervenous (Active Comparator): intravenously administrated morphine
  Interventions: Drug: intravenous morphine via PCA

INTERVENTIONS:
Drug: epidural morphine via PCEA
  Arms: morphine, epidural
Drug: epidural fentanyl via PCEA
  Arms: fentanyl, epidural
Drug: epidural methadone via PCEA
  Arms: methadone, epidural
Drug: intravenous morphine via PCA
  Arms: morphine, intervenous

SUMMARY:
The current study aim is to compare between the opioids morphine, fentanyl and methadone in terms of efficacy and side effects profile when administered epidurally for pain management after laparotomies. Intravenous morphine will also be used. The outcomes of that method will be compared to those obtained using epidurally administered opioids, as this is another commonly used postoperative pain relief method.

ELIGIBILITY:
Inclusion Criteria:

* Elective laparotomy

Exclusion Criteria:

* Subjects with diabetes mellitus, other neurological or systemic disease associated with altered sensory perception
* Illicit drug abusers
* Chronic use of pain medication
* Inability to understand consent form
* Age < 18
* Renal failure (Clcr<50 ml/min)
* Chronic use of drugs that can alter plasma levels and\or effect of the study drugs
* Corrected Q-T interval(QTc)=450msc and above
* Contra-indication for epidural catheter insertion
* Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Variable stimuli, fixed response: measurement of pain tolerance by gradual increase of temperature (quantitative sensory testing (QST))as compared to baseline | 72 hours post operatively
Fixed stimuli, variable response: measurement of reaction to fixed temperature by visual analog scale (VAS) as well as Variable stimuli, variable response (electrical stimuli)as compared to baseline. | 72 hours post operatively
patient controlled epidural analgesia (PCEI)/patient controlled analgesia (PCA)dose frequency as compared to baseline | 72 hours post operatively

SECONDARY OUTCOMES:
Measurement of opioid concentration in plasma as compared to baseline | Baseline, 4 hours post surgery and twice daily for 72 hours starting 18-24 hours post surgery
Pupillometry as compared to baseline | Baseline and twice daily for 72 hours starting 18-24 hours post surgery
Respiratory rate as compared to baseline | Baseline, 4 hours post surgery and twice daily for 72 hours starting 18-24 hours post surgery
Nasal capnography at rest as compared to baseline | Baseline and twice daily for 72 hours starting 18-24 hours post surgery
Report of adverse effects' severity as compared to baseline | Baseline, 4 hours post surgery and twice daily for 72 hours starting 18-24 hours post surgery
Report of pain severity- at rest, cough and deep breathing as compared to baseline | Baseline, 4 hours post surgery and twice daily for 72 hours starting 18-24 hours post surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel